CLINICAL TRIAL: NCT07283887
Title: Romosozumab and Denosumab, Alone or Combined, in Postmenopausal Osteoporosis: A Three-Arm Randomized Pilot Trial
Brief Title: Romosozumab and Denosumab, Alone or Combined, in Postmenopausal Osteoporosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202509047MINA
Record Dates: First submitted 2025-12-07; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis
Keywords: romosozumab; denosumab; combination therapy
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; romosozumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Denosumab (Active Comparator): After study entry, a single dose of denosumab will be administered for a six-month duration.
  Interventions: Drug: Denosumab
- Romosozumab (Active Comparator): After study entry, romosozumab will be administered monthly for six months.
  Interventions: Drug: Romosozumab
- Romosozumab plus denosumab (Experimental): After study entry, a single dose of denosumab will be administered. Romosozumab will be given monthly for six months.
  Interventions: Drug: Denosumab; Drug: Romosozumab

INTERVENTIONS:
Drug: Denosumab — After study entry, a single dose of denosumab will be administered for a six-month duration.
  Arms: Denosumab; Romosozumab plus denosumab
Drug: Romosozumab — After study entry, romosozumab will be administered monthly for six months.
  Arms: Romosozumab; Romosozumab plus denosumab

SUMMARY:
Osteoporosis is a lifelong chronic condition requiring long-term management. Conventional first-line anti-resorptive therapies often yield slow BMD improvement and may plateau after years of treatment. Recent AACE/ACE guidelines recommend anabolic agents as initial therapy in patients with severe osteoporosis or very high fracture risk; however, even anabolic monotherapy may be insufficient, with many patients failing to reach a T-score ≥ -2.5. To address this unmet need, we propose a pilot study exploring cyclic treatment using romosozumab combined with denosumab, compared with standard denosumab monotherapy. In addition to monitoring biochemical bone markers and BMD, we will incorporate imaging feature extraction from X-rays and AI-based radiomic analysis to identify imaging biomarkers that may support precision treatment strategies.

This single-center, open-label, 6-month, randomized pilot trial will enroll 90 postmenopausal women with osteoporosis (T-score ≤ -2.5) at NTUH Yunlin Branch, randomized 1:1:1 into three arms: denosumab alone, romosozumab alone, or combined therapy. The primary endpoint is percent change in lumbar spine BMD at 6 months; secondary outcomes include hip and femoral neck BMD, bone turnover markers (CTX, P1NP), fracture incidence, and adverse events. Results will estimate effect size and synergy to inform future large-scale RCTs and clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women over 50 years of age eligible for osteoporosis treatment, defined as having a bone mineral density (BMD) T-score ≤ -2.5 at the lumbar spine, total hip, or femoral neck, and who have never received osteoporosis medications (including both injectable and oral agents); or those who have used oral osteoporosis medications for no more than six months and have discontinued them for at least three months; or those who have previously received injectable osteoporosis drugs but have discontinued them for more than two years.

Exclusion Criteria:

* Age >80 years; continuous corticosteroid use; secondary osteoporosis; current use of medications affecting bone metabolism; ongoing hormone replacement therapy; metabolic bone disorders; active cancer; hypocalcemia; continued use of any osteoporosis treatment without an adequate washout period; contraindications to denosumab; and contraindications to romosozumab, such as a history of myocardial infarction or stroke within the past year.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 90 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
6-Month Percentage Change in PA Spine BMD | 6 months
  Percentage change from baseline in PA spine BMD at 6 months

SECONDARY OUTCOMES:
6-Month Percentage Change in femoral neck BMD | 6 months
  Percentage change from baseline in femoral neck BMD at 6 months
6-Month Percentage Change in total hip BMD | 6 months
  Percentage change from baseline in total hip BMD at 6 months
Percentage Change in Serum CTX at 6 Months | 6 months
  Six-month percentage change in CTX from baseline.
Percentage Change in Serum P1NP at 6 Months | 6 months
  Six-month percentage change in P1NP from baseline.

OTHER OUTCOMES:
Changes in Bone Metabolism Markers | 6 months
  Changes in OPG, RANKL, and Osteocalcin
Radiographic Changes at Hip and Spine | 6 months
  X-ray Changes in Hip, Spine, and Pelvis
Incidence of Clinical Osteoporotic Fractures | 6 months
  Clinical Osteoporotic Fracture Rate
Change in Quality of Life | 6 months
  Change in Quality of Life, measured by EQ5D5L
Safety Outcome: Adverse Events | 6 months
  any Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No